CLINICAL TRIAL: NCT04969289
Title: A Digital Intervention to Improve the Sexual and Reproductive Health of Male Adolescent Emergency Department Patients
Brief Title: A Trial of an Adolescent Male Sexual Health Intervention
Acronym: DrEric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Lauren S. Chernick, Associate Professor of Emergency Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT6680; R21NR019181 (NIH)
Record Dates: First submitted 2021-06-30; First posted 2021-07-20 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Contraception Behavior
Keywords: Digital health; Sexual health; Sexual education; Adolescent health; Mobile health
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Intervention participants receive the Dr. Eric program. Control participants will receive the standard of care.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be electronic. If assessed via phone call, outcome assessors will be blinded to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dr. Eric Digital Health Intervention (Experimental): Participants will interact with an ED-based iPad and the Dr. Eric app for a recorded period of time. After completion, an animated video will explain the ERIC texting program and "live" office hours. The participant enters his phone number and then receives a welcome text. Weekly texts are sent directly to the participant phone via short message service (SMS).
  Interventions: Behavioral: Dr. Eric Digital Health Intervention
- Standard of Care (No Intervention): Participants randomized to the SC arm will receive standard medical care as determined by the ED provider, which is typically referral to a primary care or adolescent provider. Mobile telephone numbers will be collected for follow up purposes.

INTERVENTIONS:
Behavioral: Dr. Eric Digital Health Intervention — Dr. Eric is a user-informed, theory-based, digital health intervention that aims to improve adolescent male SRH. This ED-based intervention consists of two parts-an interactive, tailored app and 3 months of personalized, two-way text messaging. It is based on an evidence-based sexual health curriculum we developed using established behavioral theories, prior literature, input from key stakeholders, qualitative patient interviews, and our prior ED-based work.
  Arms: Dr. Eric Digital Health Intervention

SUMMARY:
Early unintended fatherhood and rates of sexually transmitted infections remain national concerns, disproportionately affecting minority, underserved adolescent males, many of whom frequently use emergency departments (EDs) for medical care. EDs must implement effective sexual and reproductive health interventions that are evidence-based and reproducible. This research will conduct pilot testing of a personalized and interactive digital intervention specifically targeting adolescent males entitled Dr. Eric that is theory-based, user-informed, and scalable across EDs.

DETAILED DESCRIPTION:
Emergency Departments (EDs) care for 19 million adolescents each year, the majority of whom are low-income, racial and ethnic minorities, and participating in risky sexual behaviors. Despite a growing interest in expanding the role of the ED to provide preventive care, ED providers identify limited resources and time constraints as barriers to the implementation of public health interventions. Novel interventions are needed that fit efficiently within the ED workflow. The prior work of these investigators highlighted a significant public health problem-high risk sex among the adolescent male ED population. The investigators demonstrated that adolescent male ED patients are frequently having sex without condoms, increasing their risk of unintended early fatherhood and sexually transmitted infections (STI). These adolescents admit to low knowledge of effective contraceptive methods and having few discussions with medical providers and sexual partners about these methods. However, these male adolescents are receptive to sexual and reproductive health (SRH) interventions, particularly during the ED visit and via digital technology. They are particularly interested in interventions that feel relatable and are from a trustworthy source. To date, no intervention has successfully increased contraceptive use among this high risk, hard-to-reach ED population. Additionally, although evidence suggests that SRH digital interventions can improve SRH health, few interventions specifically target males. To improve adolescent SRH outcomes, the investigators have gathered an accomplished team with expertise in adolescent health, ED-based clinical trials, mobile health, and user-informed digital interventions. They created a novel intervention of an ED-based, theory-based, user-informed SRH digital intervention that includes a tailored educational app and 3 months of personalized and interactive text messaging. In this study, the investigators will conduct a pilot randomized controlled trial of Dr. Eric (Emergency Room Interventions to improve Care) to assess implementation outcomes and potential effectiveness. The investigators hypothesize that the Dr. Eric intervention will be feasible in the ED setting, be acceptable to adolescent males, demonstrate fidelity, and be adopted by users. The investigators also hypothesize that sexually active adolescent male ED patients who receive Dr. Eric will more often have consistent condom use than those who receive standard outpatient referral alone. These data will inform a subsequent multi-center clinical trial with sufficient power to measure clinically significant changes in consistent condom use. Ultimately, a digital ED-based intervention that is effective and automated can be utilized by other EDs as a reproducible and scalable means to promote sexual and reproductive preventive care, decrease unintended early fatherhood and STI risk among adolescent males, and improve adolescent health outcomes throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* ED male adolescent patients aged 14-21 years
* sexually active (vaginal intercourse) with females in the past 3 months

Exclusion Criteria:

* do not own a mobile phone
* too ill per the attending
* are cognitively impaired
* does not speak English
* want their partner to become pregnant in the next year

Ages: 14 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 119 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Chernick, MD MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic and behavioral data from baseline questionnaires, telephone follow up, and text message data collection. It will also contain usability testing information. All participants will be assigned a unique identifier and all data will remain confidential.
Time Frame: Data will become available after study analysis is completed, at least one year after study completion.
Access Criteria: Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2021 to June 2022, 119 male participants were enrolled and randomized.
Pre-assignment Details: The investigators excluded 9 patients in the intervention arm and 13 patients from the standard control arm in the analysis as they were lost to follow-up.
Period: Overall Study
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
Started | 60 | 59
Completed | 47 | 50
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 13 | 9

BASELINE CHARACTERISTICS:
Population: We enrolled 60 in the intervention and 59 in the control arm.
Groups:
- Dr. Eric Digital Health Intervention: Dr. Eric Digital Health Intervention: Dr. Eric is a user-informed, theory-based, digital health intervention that aims to improve adolescent male sexula health. This ED-based intervention consists of two parts-an interactive, tailored app and 3 months of personalized, two-way text messaging. It is based on an evidence-based sexual health curriculum we developed using established behavioral theories, prior literature, input from key stakeholders, qualitative patient interviews, and our prior ED-based work.
- Total: Total of all reporting groups
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 35 | 77
  Between 18 and 65 years | 18 | 24 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 59 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 47 | 92
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119
Condom use at last intercourse [Count of Participants; unit: Participants] | 36 | 26 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Participants Who Agreed to be Enrolled in the Study
Description: Implementation, feasibility: This outcome is designed to measure feasibility - the extent to which an innovation can be used in a setting. The investigators will measure the number of participants who are eligible, and agree to be enrolled into the study.
Time Frame: From day 1 of enrollment until the final day of enrollment (1 year)
Measure: Number; unit: participants
Groups:
- All Eligible Patients: All eligible male patients aged 14-21 assessed for screening and eligible for enrollment
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 138
participants | 119

2. Primary Outcome: Number of Participants That Are Lost to Follow up (at Each Time Point)
Description: Implementation, feasibility: This outcome is to measure feasibility for both arms in which feasibility is defined as the extent to which an innovation can be used in a setting. The investigators will measure the number of participants in each arm that are lost to follow up in each respective arm at the 6 and 13 week time point. Lost to follow up means that we tried to contact the participant to assess outcome measures but they did not respond to texts or phone calls.
Time Frame: 6 and 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
Number analyzed (Participants) | 60 | 59
Participants
  6 weeks | 25 | 13
  13 weeks | 19 | 13

3. Primary Outcome: Total Number of Participants Who Demonstrated Acceptability (Intervention Arm ONLY)
Description: Implementation, acceptability: This outcome is to measure acceptability for the intervention group only. Acceptability is the extent to which the innovation is agreeable to a stakeholder. The investigators asked the Agree/Disagree question of "Dr. Eric meets my approval," as self-reported after app completion.
Time Frame: From day 1 of enrollment until the final day of enrollment (1 year)
Population: Only includes participants from this intervention arm.
Measure: Number; unit: participants
Groups:
- Intervention Participants: Those in the intervention arm
Arm/Group | Intervention Participants
Number analyzed (Participants) | 60
participants | 53

4. Primary Outcome: The Number of Participants Who Interacted With All 5 Educational Modules (Intervention Arm ONLY)
Description: Implementation, adoption: This outcome is for the intervention group only. Th investigators assessed adoption by measuring the number of intervention participants who interacted with all 5 educational modules, based off of data that is recorded by the app.
Time Frame: From day 1 of enrollment until the final day of enrollment (1 year)
Population: Only includes participants from this intervention arm.
Measure: Number; unit: participants
Groups:
- Intervention Arm: Those in the intervention arm
Arm/Group | Intervention Arm
Number analyzed (Participants) | 60
participants | 59

5. Primary Outcome: Number of Participants Who Opt Out of the Texting Messaging Component of the Program (Intervention Arm ONLY)
Description: Implementation, fidelity: This outcome is for the intervention group only. Fidelity is the extent to which an intervention is used as intended. This outcome measures the number of participants in the intervention group who opt out of the texting messaging component of the program.
Time Frame: 3 months
Population: Only includes participants from this intervention arm.
Measure: Number; unit: participants who opted out of texting
Arm/Group | Intervention Arm
Number analyzed (Participants) | 60
participants who opted out of texting | 14

6. Primary Outcome: Percentage of Condom Use Among Participants
Description: Efficacy, Consistent Condom Use: This outcome is designed to measure efficacy and is a self-reported outcome and only includes participants who completed follow-up at 13 weeks. Percentages are calculated by dividing the total number of episodes of vaginal intercourse by the total number of times a male condom was used during vaginal intercourse over the past 4 weeks to report percentage of condom use within each arm.
Time Frame: 3 months (or 13 weeks)
Population: Calculated from participants who completed follow-up at 13 weeks.
Measure: Number; unit: percentage of episodes of condom-sex
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
Number analyzed (Participants) | 41 | 46
percentage of episodes of condom-sex | 34.6 | 37.3

7. Primary Outcome: Percentage of Condom Use Among Participants
Description: Efficacy, Consistent Condom Use: This outcome is designed to measure efficacy and is a self-reported outcome. This outcome only includes participants who completed follow-up at 6 weeks and were sexually active in the prior 4 weeks. The percentages are calculated by dividing the total number of episodes of vaginal intercourse by the total number of times a male condom was used during vaginal intercourse over the past 4 weeks to report percentages of condom use within each arm.
Time Frame: 6 weeks
Population: Includes participants who completed follow-up at 6 weeks and were sexually active in the prior 4 weeks.
Measure: Number; unit: percentage of episodes of condom-sex
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
Number analyzed (Participants) | 23 | 28
percentage of episodes of condom-sex | 82.5 | 47.5

8. Secondary Outcome: Number of Participants Who Had Intercourse Over the Past 4 Weeks
Description: Efficacy, Abstinent: This outcome is self-reported where participants are asked if they had penile-vaginal intercourse over the past 4 week. The binary outcome is measured from a "Yes" or "No" response.
Time Frame: 3 month (13 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Participants Who Completed 3 Month Follow-up Questions; Control Participants Who Completed 3 Month Follow-up Questions: This number refers to those who completed the follow-up survey in completion which included secondary outcomes.
Arm/Group | Intervention Participants Who Completed 3 Month Follow-up Questions | Control Participants Who Completed 3 Month Follow-up Questions
Number analyzed (Participants) | 41 | 46
Participants | 5 | 9

9. Secondary Outcome: Number of Participants Who Talked to a Partner About Ways to Prevent Pregnancy Over the Past 3 Months
Description: Efficacy, Talked to a partner about ways to prevent pregnancy over the past 3 months: This outcome is based on self-reported responses on the follow-up survey in which the binary outcome is measured from a "Yes" or "No" response.
Time Frame: 3 month (13 weeks)
Population: This count only includes participants who completed this question in the follow-up survey.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Participants Who Completed 3 Month Follow-up Questions; Control Participants Who Completed 3 Month Follow-up Questions: This number refers to those who completed this question in the follow-up survey.
Arm/Group | Intervention Participants Who Completed 3 Month Follow-up Questions | Control Participants Who Completed 3 Month Follow-up Questions
Number analyzed (Participants) | 36 | 46
Participants | 23 | 29

10. Secondary Outcome: Number of Participants Who Tested for a Sexually Transmitted Infection Over the Past 3 Months
Description: Efficacy, Tested for a sexually transmitted infection over the past 3 months: This outcome is based on self-reported responses on the follow-up survey, in which the binary outcome is measured from a "Yes" or "No" response.
Time Frame: 3 month (13 weeks)
Population: Only includes participants who completed this question in the follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Participants Who Completed 3 Month Follow-up Questions | Control Participants Who Completed 3 Month Follow-up Questions
Number analyzed (Participants) | 42 | 46
Participants | 13 | 15

11. Secondary Outcome: Number of Participants Who Tested for HIV Over the Past 3 Months
Description: Efficacy, Tested for HIV over the past 3 months: This outcome was based on self-reported responses on the follow-up survey in which the binary outcome is measured from a "Yes" or "No" response.
Time Frame: 3 month (13 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Participants Who Completed 3 Month Follow-up Questions | Control Participants Who Completed 3 Month Follow-up Questions
Number analyzed (Participants) | 41 | 46
Participants | 9 | 15

12. Secondary Outcome: Number of Participants Who Consistently Used Condoms at Every Intercourse
Description: Efficacy, Consistent Condom Use at Every Intercourse: This outcome is designed to measure efficacy, is a self-reported outcome and only includes participants who completed follow-up at 13 weeks. Answere are binary (yes/no) to using a condom at every intercourse over the past 3 months.
Time Frame: 3 months (or 13 weeks)
Population: Calculated from participants who completed follow-up at 13 weeks and were sexually active in the past 3 months.
Measure: Number; unit: participants
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
Number analyzed (Participants) | 26 | 24
participants | 12 | 13

13. Secondary Outcome: Number of Participants Who Used a Condom at Last Intercourse
Description: Efficacy, Use a condom at last intercourse: This outcome is designed to measure efficacy, is a self-reported outcome and only includes participants who completed follow-up at 13 weeks and were sexually active. Answers are binary (yes/no) to the question if a condom was used at last intercourse.
Time Frame: 3 months (or 13 weeks)
Population: Calculated from participants who completed follow-up at 13 weeks and were sexually active.
Measure: Number; unit: participants
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
Number analyzed (Participants) | 26 | 24
participants | 18 | 20

14. Secondary Outcome: Number of Participants Who Used Any Contraceptive Method at Last Intercourse
Description: Efficacy, Used any method of contraception at last intercourse: This outcome is based on self-reported responses on the follow-up survey in which the binary outcome is measured from a "Yes" or "No" response.
Time Frame: 3 month (13 weeks)
Population: Only includes participants who completed this question in the follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Participants Who Completed 3 Month Follow-up Questions | Control Participants Who Completed 3 Month Follow-up Questions
Number analyzed (Participants) | 26 | 24
Participants | 22 | 20

ADVERSE EVENTS:
Time Frame: From the date of the first enrollment to the date of the final assessment of outcome measures (1 year and 3 months)
Description: We defined an Adverse Event as an event where a participant felt threatened or is hurt due to the Dr. Eric intervention. This is a question we ask in our follow-up survey.
Arm/Group | Dr. Eric Digital Health Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/59

LIMITATIONS AND CAVEATS:
This study included individuals who predominately identified as Hispanic and "more than one race"; the investigators did not ask for more granular race and ethnicity data. Also, the investigators were limited in their ability to assess additional measures of adoption and fidelity such as time spent on the app, which would have represented real use. For the primary outcome, the investigators measured condom use as a group; different results could occur if they measured use by person.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04969289/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04969289/ICF_001.pdf